CLINICAL TRIAL: NCT06558292
Title: The Effect of a Pre-Clinical Practice Simulation Using Virtual Reality Stress and Anxiety Levels Among Nursing Students on Operating Room: A Randomised Controlled Trial
Brief Title: The Effect of a Pre-Clinical Practice Simulation Using Virtual Reality Stress and Anxiety Levels
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Emine Arici Parlak, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14141414
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Clinical Practice; Virtual Reality; Nursing Education; Nursing Students; Simulation
Keywords: Clinical practice; Virtual Reality; Nursing Students; Simulation; Stress; Anxiety; Operating Room
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Students will experience the operating room environment with virtual reality glasses before clinical practice.
  Anxiety and stress will be evaluated in clinical practice
  Interventions: Other: Virtual Reality Group
- Control Group (No Intervention): Anxiety and stress will be evaluated in clinical practice

INTERVENTIONS:
Other: Virtual Reality Group — Students will experience the operating room environment with virtual reality glasses before clinical practice.
  Arms: Virtual Reality Group

SUMMARY:
This study is designed as a randomized controlled trial to examine the effect of simulation practices using virtual reality headsets related to the operating room environment on nursing students' stress and anxiety levels before clinical practice.

DETAILED DESCRIPTION:
Nursing education is a field that requires the integration of both clinical and theoretical training, as it is a practical discipline (Ryan et al., 2010; Özçelik & Ayhan, 2021). Therefore, nurse educators must continuously innovate their teaching and learning methods at every stage of their students' educational journey (Fealy et al., 2019). The use of simulation in nursing education has been implemented for the past 50 years (Foronda et al., 2017). Simulation practices can reflect the characteristics of the real world, providing students with safe learning environments where they can practice until they achieve skill competence through feedback and self-correction (Aebersold, 2018; Shorey & Ng, 2021). With the advancement of simulation technology over time, it is observed that the realism and authenticity of simulated environments have increased.

Upon reviewing the literature, no studies were found that evaluate the impact of simulation practices using virtual reality headsets related to the operating room environment on nursing students' stress and anxiety levels before clinical practice. Therefore, this study is planned to be conducted on nursing students. The results of this study are expected to contribute to educators in enhancing, planning, and managing the effectiveness of clinical education.

The study will conduct as a prospective randomized controlled trial. After obtaining verbal and written consent from the students before and after the clinical practice, the study will conduct with various data collection forms.

These forms are; Student Identification form, Spielberger's State and Trait Anxiety Inventory, Student Satisfaction and Self-Confidence in Learning Scale and Perceived Stress Scale for Nursing Students will be used, and Visual Analog Scale will be used to assess the general self-confidence of the students. Patients will randomize.

The Virtual Reality (VR) group in group- I (n=41), and group II (n=41) will be the control group. We have three stage. In first stage; anxiety levels will be measured for both groups. In second stage; Student Satisfaction and Self-Confidence in Learning Scale and anxiety levels will evaluated for the Virtual Reality (VR) group in group- I. In third stage; anxiety levels and Stress levels will be measured for both groups in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Being a second-year student at Gülhane Nursing Faculty of Health Sciences University
* Agreeing to participate in the study

Exclusion Criteria:

* Not completing any stage of the study
* Wanting to withdraw from the study
* Having previously taken the surgical disease nursing course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Having taken a course in surgical diseases nursing
Enrollment: 82 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from anxiety and stress level in clinical practice | After Simulation Using Virtual Reality in clinical pratice. An average of 1 year.
  The simulation application of the operating room environment with virtual reality glasses to nursing students before clinical practice will affect the stress and anxiety levels of the students in the operating room. This status will evaluate with Spielberger's State and Trait Anxiety Inventory and Perceived Stress Scale for Nursing Students Spielberger's State and Trait Anxiety Inventory consists of a total of 40 items, 20 for each scale. The first form in the inventory includes statements about state anxiety, and the second form includes statements about trait anxiety High scores indicate high anxiety levels. Perceived Stress Scale for Nursing Students consists of 29 items and 6 sub-dimensions. Total score is 0-116 (sub-dimension total scores are: 0-12, 0-32, 0-20, 0-24, 0-12, 0-16). Higher scores indicate higher levels of stress. (Sheu et al. 2002).

SECONDARY OUTCOMES:
Change from confidence level in clinical practice | After Simulation Using Virtual Reality in clinical pratice. An average of 1 year
  In this section, the degree of confidence level will increase or not decrease . This status will evaluate with Visual Analogue Scale (VAS). VAS is a horizontal line with a length of 10 cm. According to VAS, 0 is the lowest level and 10 is the highest level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkiye Gulhane Faculty of Nursing, Ankara, Turkey (Türkiye)